CLINICAL TRIAL: NCT02391116
Title: An Open-label, Single-arm Phase II Study in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL) to Evaluate Efficacy and Safety of Treatment With Single Agent Copanlisib and the Impact of Biomarkers Thereupon.
Brief Title: Phase II Copanlisib in Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17119; 2014-004848-36 (EudraCT Number)
Record Dates: First submitted 2015-02-16; First posted 2015-03-18 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib (Aliqopa, BAY80-6946) (Experimental): Copanlisib (Aliqopa, BAY80-6946) solution for IV infusion (test drug/investigational medicinal product)
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — Participants assigned to receive copanlisib intravenous (IV) infusion at a dose of 60 mg as single agent on Days 1, 8, and 15 of 28-day treatment cycle. Copanlisib treatment was to be continued until disease progression (PD), unacceptable toxicity, or until another criterion was met for withdrawal from the study treatment

SUMMARY:
To assess the potential efficacy (in terms of objective response) of single agent copanlisib in patients with relapsed or refractory Diffuse large B-cell lymphoma (DLBCL) and assess the relationship between efficacy and a potentially predictive biomarker

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diffuse large B-cell lymphoma (DLBCL) (de novo or DLBCL transformed from follicular lymphoma on the basis of a tissue biopsy).
* Received at least one prior therapy for aggressive Non-Hodgkin's Lymphoma (NHL) (DLBCL).
* Received CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone) + rituximab or equivalent regimen.
* Patients must have measurable disease.
* Not eligible or not willing to receive the high-dose (myeloablative) chemotherapy (HDC) and stem cell transplant (SCT).
* A fresh tumor biopsy collected during screening and /or archival tumor tissue collected after the last relapse/disease progression.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
* Left ventricular ejection fraction (LVEF) ≥ the lower limit of normal (LLN) for the Institution. (as per local standard of care) as measured by echocardiogram (ECHO) or Multiple gated acquisition (MUGA) scan.
* Adequate bone marrow, liver and renal function.

Exclusion Criteria:

* Any of the following as the only site(s) of disease: palpable lymph nodes not visible on imaging studies, skin lesions, or bone marrow involvement only.
* Active CTCAE (Common Terminology Criteria for Adverse Events) Grade 3/4 infection.
* Current central nervous system (CNS) involvement by lymphoma.
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction within the past 6 months before start of study treatment.
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion).
* Type I or II diabetes mellitus with HbA1c > 8.5% at Screening.
* New York Heart Association (NYHA) class III or IV heart disease.
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator).
* Patients who previously received therapy with copanlisib or other PI3K inhibitors are not eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (30):
- Australia (4):
  - Kingswood, New South Wales
  - Ballarat, Victoria
  - Prahran, Victoria
  - Box Hill
- Belgium (5):
  - Wilrijk, Antwerpen
  - Bruxelles - Brussel
  - Edegem
  - Ghent
  - Leuven
- Canada (4):
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Denmark (2):
  - Aarhus C
  - Odense C
- France (6):
  - Caen
  - Créteil
  - Lille
  - Paris
  - Pierre-Bénite
  - Poitiers
- Germany (3):
  - Münster, North Rhine-Westphalia
  - Leipzig, Saxony
  - Berlin
- Milan, Lombardy, Italy
- Singapore, Singapore
- Seoul, South Korea
- United Kingdom (3):
  - Truro, Cornwall
  - Southampton, Hampshire
  - London

REFERENCES:
- [Derived] Lenz G, Hawkes E, Verhoef G, Haioun C, Thye Lim S, Seog Heo D, Ardeshna K, Chong G, Haaber J, Shi W, Gorbatchevsky I, Lippert S, Hiemeyer F, Piraino P, Beckmann G, Pena C, Buvaylo V, Childs BH, Salles G. Single-agent activity of phosphatidylinositol 3-kinase inhibition with copanlisib in patients with molecularly defined relapsed or refractory diffuse large B-cell lymphoma. Leukemia. 2020 Aug;34(8):2184-2197. doi: 10.1038/s41375-020-0743-y. Epub 2020 Feb 14. PMID 32060403
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 centers across 10 countries, between 08 May 2015 (first patient first visit) and 18 January 2018 (last patient last visit).
Pre-assignment Details: A total of 91 participants were screened, of which 67 were assigned to study treatment and also started the treatment, and 24 were screened but never assigned to treatment. Altogether 27 participants were excluded from the per protocol set, which comprised 40 participants.
Period: Treatment
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Started | 67
Included in Per Protocol Set | 40
Completed | 53 (Reasons for completion in this period included death (2), PD (50) and lack of efficacy (1))
Not Completed | 14
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Adverse Event (AE) Without Clinical PD | 9
Not completed — AE with Clinical PD | 3
Period: Safety Follow-up
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Started | 56 (This period excludes 2 deaths on treatment and 9 participants entering active follow-up)
Completed | 43 (14 participants were considered completed due to death)
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4
Not completed — Switching to Other Therapy | 4
Not completed — No Follow Up | 1
Not completed — Deterioration of General Conditions | 3
Period: Active Follow-up
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Started | 9 (This period incorporates safety follow-up with radiological)
Completed | 6 (Reasons for completion in this period included death (2) and PD (4))
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Switching to Other Therapy | 2
Period: Survival Follow-up
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Started | 46 (21 participants discontinued from treatment didn't enter due to withdrawal by subject (3) and death)
Completed | 42 (Reason for completed in this period included death (35) and clinical endpoint reached (7))
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Switching to Other Therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full analysis set (FAS) and per protocol set (PPS)
  Years
    Full analysis set (FAS) | 65.3 (14.5)
    Per protocol set (PPS): number analyzed (Participants) | 40
    Per protocol set (PPS) | 69.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set (FAS) and per protocol set (PPS)
  Participants
    Full analysis set (FAS): Female | 28
    Full analysis set (FAS): Male | 39
    Per protocol set (PPS): number analyzed (Participants) | 40
    Per protocol set (PPS): Female | 15
    Per protocol set (PPS): Male | 25
CD79b Status [Count of Participants; unit: Participants] — Population: Full analysis set (FAS) and per protocol set (PPS)
  Participants
    Full analysis set (FAS): CD79b Mutant | 9
    Full analysis set (FAS): CD79b Wild-type | 45
    Full analysis set (FAS): CD79b Status Missing | 13
    Per protocol set (PPS): number analyzed (Participants) | 40
    Per protocol set (PPS): CD79b Mutant | 8
    Per protocol set (PPS): CD79b Wild-type | 32
    Per protocol set (PPS): CD79b Status Missing | 0
DLBCL / Cell of Origin (COO) Subtype [Count of Participants; unit: Participants] — Population: Full analysis set (FAS) and per protocol set (PPS)
  Participants
    Full analysis set (FAS): Activated B-cell-like (ABC) | 19
    Full analysis set (FAS): Germinal center B-cell-like (GCB) | 30
    Full analysis set (FAS): Unclassifiable | 3
    Full analysis set (FAS): DLBCL/COO Subtype Missing | 15
    Per protocol set (PPS): number analyzed (Participants) | 40
    Per protocol set (PPS): Activated B-cell-like (ABC) | 16
    Per protocol set (PPS): Germinal center B-cell-like (GCB) | 22
    Per protocol set (PPS): Unclassifiable | 2
    Per protocol set (PPS): DLBCL/COO Subtype Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Total Population Based on Investigator Assessment
Description: The objective response rate (ORR) was defined as the percentage of participants who had at least one post-baseline overall response of complete response (CR) or partial response (PR) during study conduct according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT. The primary efficacy overall response assessment was based on investigator assessment of response.
Time Frame: From start of study treatment assessed up to 24 weeks after the last participant fully evaluable for the primary endpoint started treatment (about 12 months)
Population: Full analysis set (FAS) and per protocol set (PPS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Percentage of participants
  Full analysis set (FAS) | 19.4 [11.9 to 29.1]
  Per protocol set (PPS): number analyzed (Participants) | 40
  Per protocol set (PPS) | 25.0 [14.2 to 38.7]

2. Primary Outcome: ORR by CD79b Status Based on Investigator Assessment
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full analysis set (FAS) and per protocol set (PPS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- CD79b Mutant: Included all participants with CD79b mutant classified at baseline depending on the biomarker value
- CD79b Wild-type: Included all participants with CD79b wild-type classified at baseline depending on biomarker value
- CD79b Status Missing: Included all participants with CD79b status missing at baseline
Arm/Group | CD79b Mutant | CD79b Wild-type | CD79b Status Missing
Number analyzed (Participants) | 9 | 45 | 13
Percentage of participants
  Full analysis set (FAS) | 22.2 [4.1 to 55.0] | 20.0 [10.9 to 32.3] | 15.4 [2.8 to 41.0]
  Per protocol set (PPS): number analyzed (Participants) | 8 | 32 | 0
  Per protocol set (PPS) | 25.0 [4.6 to 60.0] | 25.0 [13.1 to 40.6] |
Statistical Analysis 1: Comparison: CD79b Mutant vs CD79b Wild-type; Test type: Other; Exact confidence intervals (CI); Percentage Difference = 2.2, 90% CI 2-sided [-28.7 to 32.9] — ORR difference in FAS (N=54): ORR in CD79b mutant subgroup minus ORR in CD79b wild-type subgroup
Statistical Analysis 2: Comparison: CD79b Mutant vs CD79b Wild-type; Test type: Other; Exact confidence intervals (CI); Percentage Difference = 0.0, 90% CI 2-sided [-33.5 to 33.5] — ORR difference in PPS (N=40): ORR in CD79b mutant subgroup minus ORR in CD79b wild-type subgroup

3. Primary Outcome: ORR by DLBCL/COO Subtype Based on Investigator Assessment
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full analysis set (FAS) and per protocol set (PPS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Activated B-cell-like (ABC): Included all participants with activated B-cell-like (ABC) DLBCL classified at baseline depending on the biomarker value
- Germinal Center B-cell-like (GCB): Included all participants with germinal center B-cell-like (GCB) DLBCL classified at baseline depending on the biomarker value
- Unclassifiable: Included all participants with unclassifiable DLBCL/COO subtype at baseline
- DLBCL/COO Subtype Missing: Included all participants with DLBCL/COO subtype missing at baseline
Arm/Group | Activated B-cell-like (ABC) | Germinal Center B-cell-like (GCB) | Unclassifiable | DLBCL/COO Subtype Missing
Number analyzed (Participants) | 19 | 30 | 3 | 15
Percentage of participants
  Full analysis set (FAS) | 31.6 [14.7 to 53.0] | 13.3 [4.7 to 28.0] | 33.3 [1.7 to 86.5] | 13.3 [2.4 to 36.3]
  Per protocol set (PPS): number analyzed (Participants) | 16 | 22 | 2 | 0
  Per protocol set (PPS) | 37.5 [17.8 to 60.9] | 13.6 [3.8 to 31.6] | 50.0 [2.5 to 97.5] |
Statistical Analysis 1: Comparison: Activated B-cell-like (ABC) vs Germinal Center B-cell-like (GCB) vs Unclassifiable; Test type: Other; Exact confidence intervals (CI); Percentage Difference = 16.4, 90% CI 2-sided [-7.2 to 39.1] — ORR difference in FAS (N=52): ORR in ABC subgroup minus ORR in non-ABC group (i.e. combined GCB subgroup and Unclassifiable subgroup)
Statistical Analysis 2: Comparison: Activated B-cell-like (ABC) vs Germinal Center B-cell-like (GCB) vs Unclassifiable; Test type: Other; Exact confidence intervals (CI); Percentage Difference = 20.8, 90% CI 2-sided [-6.8 to 46.2] — ORR difference in PPS (N=40): ORR in ABC subgroup minus ORR in non-ABC group (i.e. combined GCB subgroup and Unclassifiable subgroup)
Statistical Analysis 3: Comparison: Activated B-cell-like (ABC) vs Germinal Center B-cell-like (GCB) vs Unclassifiable; Test type: Other; Exact confidence intervals (CI); Percentage Difference = -18.5, 90% CI 2-sided [-40.1 to 4.6] — ORR difference in FAS (N=52): ORR in GCB subgroup minus ORR in non-GCB subgroup (i.e. combined ABC subgroup and Unclassifiable subgroup)
Statistical Analysis 4: Comparison: Activated B-cell-like (ABC) vs Germinal Center B-cell-like (GCB) vs Unclassifiable; Test type: Other; Exact confidence intervals (CI); Percentage Difference = -25.3, 90% CI 2-sided [-49.1 to 1.1] — ORR difference in PPS (N=40): ORR in GCB subgroup minus ORR in non-GCB subgroup (i.e. combined ABC subgroup and Unclassifiable subgroup)
Statistical Analysis 5: Comparison: Activated B-cell-like (ABC) vs Germinal Center B-cell-like (GCB) vs Unclassifiable; Test type: Other; Exact confidence intervals (CI); Percentage Difference = 12.9, 90% CI 2-sided [-42.4 to 63.2] — ORR difference in FAS (N=52): ORR in Unclassifiable subgroup minus ORR in ABC / GCB subgroup (i.e. combined ABC subgroup and GCB subgroup)
Statistical Analysis 6: Comparison: Activated B-cell-like (ABC) vs Germinal Center B-cell-like (GCB) vs Unclassifiable; Test type: Other; Exact confidence intervals (CI); Percentage Difference = 26.3, 90% CI 2-sided [-44.3 to 77.6] — ORR difference in PPS (N=40): ORR in Unclassifiable subgroup minus ORR in ABC / GCB subgroup (i.e. combined ABC subgroup and GCB subgroup)

4. Secondary Outcome: Duration of Response (DOR) in Total Population
Description: The duration of response (DOR) was defined as the time from the date of first observed overall response (CR or PR) until radiological PD or death due to any cause, whichever was earlier. DOR was defined for responders only (i.e. participants with a best response of CR or PR), based on the investigator assessment of tumor response according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT.
Time Frame: From start of study treatment assessed up to 2 years after the last participant's first treatment or the last participant dies, whichever occurs first
Population: Responders (i.e. participants with a best response of CR or PR) in full analysis set based on the investigator assessment
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 13
Days | 132 [57 to 345]

5. Secondary Outcome: DOR by CD79b Status
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD79b Mutant | CD79b Wild-type | CD79b Status Missing
Number analyzed (Participants) | 2 | 9 | 2
Days | 516 [417 to 615] | 113 [39 to 272] | 113 [93 to 132]

6. Secondary Outcome: DOR by DLBCL/COO Subtype
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Activated B-cell-like (ABC) | Germinal Center B-cell-like (GCB) | Unclassifiable | DLBCL/COO Subtype Missing
Number analyzed (Participants) | 6 | 4 | 1 | 2
Days | 193 [39 to 417] | 183 [63 to 615] | 52 [NA to NA] — Value cannot be estimated due to censored data. | 113 [93 to 132]

7. Secondary Outcome: Progression-free Survival (PFS) in Total Population
Description: The progression-free survival (PFS) was defined as the time from date of start of study treatment to radiological PD or death due to any cause, whichever was earlier, based on the investigator assessment of tumor response according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT.
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Days | 54 [50 to 84]

8. Secondary Outcome: PFS by CD79b Status
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD79b Mutant | CD79b Wild-type | CD79b Status Missing
Number analyzed (Participants) | 9 | 45 | 13
Days | 73 [43 to 465] | 52 [46 to 88] | 56 [46 to 138]

9. Secondary Outcome: PFS by DLBCL/COO Subtype
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Activated B-cell-like (ABC) | Germinal Center B-cell-like (GCB) | Unclassifiable | DLBCL/COO Subtype Missing
Number analyzed (Participants) | 19 | 30 | 3 | 15
Days | 73 [44 to 101] | 52 [46 to 116] | 84 [26 to 164] | 51 [33 to 58]

10. Secondary Outcome: Overall Survival (OS) in Total Population
Description: The overall survival (OS) was defined as the time from date of start of study treatment until death from any cause.
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Days | 224 [104 to 327]

11. Secondary Outcome: OS by CD79b Status
Description: The overall survival (OS) was defined as the time from date of start of study treatment until death from any cause.
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CD79b Mutant | CD79b Wild-type | CD79b Status Missing
Number analyzed (Participants) | 9 | 45 | 13
Days | 178 [57 to NA] — Value cannot be estimated due to censored data. | 242 [73 to 385] | 224 [56 to 388]

12. Secondary Outcome: OS by DLBCL/COO Subtype
Description: The overall survival (OS) was defined as the time from date of start of study treatment until death from any cause.
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Activated B-cell-like (ABC) | Germinal Center B-cell-like (GCB) | Unclassifiable | DLBCL/COO Subtype Missing
Number analyzed (Participants) | 19 | 30 | 3 | 15
Days | 210 [63 to 421] | 287 [94 to 436] | 164 [93 to 273] | 160 [46 to 400]

13. Secondary Outcome: Duration of Stable Disease (DOSD) in Total Population
Description: The duration of stable disease (DOSD) was defined as the time (in days) from date of start of study treatment to radiological PD or death due to any cause, whichever was earlier. The DOSD was only evaluated in participants failing to achieve a best response of CR or PR, but who achieved SD (stable disease), based on the investigator assessment of tumor response according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT.
Time Frame: as for outcome 4
Population: Participants who failed to achieve CR or PR but achieved SD in full analysis set based on the investigator assessment
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 14
Days | 106 [73 to 138]

14. Secondary Outcome: Disease Control Rate (DCR) in Total Population
Description: The disease control rate (DCR) was defined as the percentage of participants who had a best response rating of CR, PR, or SD that was achieved during treatment or within 30 days after termination of study drug. The tumor response was based on investigator assessment according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT.
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Percentage of participants | 40.3 [30.2 to 51.1]

15. Secondary Outcome: DCR by CD79b Status
Description: as for outcome 14
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | CD79b Mutant | CD79b Wild-type | CD79b Status Missing
Number analyzed (Participants) | 9 | 45 | 13
Percentage of participants | 55.6 [25.1 to 83.1] | 40.0 [27.7 to 53.3] | 30.8 [11.3 to 57.3]

16. Secondary Outcome: DCR by DLBCL/COO Subtype
Description: as for outcome 14
Time Frame: as for outcome 4
Population: Full analysis set (FAS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Activated B-cell-like (ABC) | Germinal Center B-cell-like (GCB) | Unclassifiable | DLBCL/COO Subtype Missing
Number analyzed (Participants) | 19 | 30 | 3 | 15
Percentage of participants | 52.6 [32.0 to 72.6] | 40.0 [25.0 to 56.6] | 33.3 [1.7 to 86.5] | 26.7 [9.7 to 51.1]

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: A TEAE was defined as any event arising or worsening after the start of study drug administration until 30 days after the last application.
Time Frame: From start of test drug to 30 days after the last test drug intake, assessed up to 2 years after the last participant's first treatment or the last participant dies (whichever occurs first), with an average of 15 weeks for individual participant
Population: Safety analysis set (SAF)
Measure: Number; unit: Participants
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Participants
  Any TEAE | 65
  Any TESAE | 44

18. Other Pre Specified Outcome: Time to Response (TTR) in Total Population
Description: The time to response (TTR) was defined as the time (days) from start of study treatment to the date of first observed response (first measured CR or PR). TTR was defined for responders only (i.e. participants with CR or PR), based on the investigator assessment of tumor response according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 13
Days | 52 [49 to 56]

19. Other Pre Specified Outcome: ORR in Total Population Based on Central Imaging Review
Description: The objective response rate (ORR) was defined as the percentage of participants who had at least one post-baseline overall response of complete response (CR) or partial response (PR) during study conduct according to the criteria defined by the Lugano Classification, 2014 and assessed by CT/MRI/PET-CT. The overall response assessment for this outcome measure was based on central imaging review.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
Number analyzed (Participants) | 67
Percentage of participants | 22.4 [14.3 to 32.4]

20. Other Pre Specified Outcome: ORR by CD79b Status Based on Central Imaging Review
Description: as for outcome 19
Time Frame: as for outcome 1
Population: Full analysis set (FAS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | CD79b Mutant | CD79b Wild-type | CD79b Status Missing
Number analyzed (Participants) | 9 | 45 | 13
Percentage of participants | 44.4 [16.9 to 74.9] | 20.0 [10.9 to 32.3] | 15.4 [2.8 to 41.0]

21. Other Pre Specified Outcome: ORR by DLBCL/COO Subtype Based on Central Imaging Review
Description: as for outcome 19
Time Frame: as for outcome 1
Population: Full analysis set (FAS)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Activated B-cell-like (ABC) | Germinal Center B-cell-like (GCB) | Unclassifiable | DLBCL/COO Subtype Missing
Number analyzed (Participants) | 19 | 30 | 3 | 15
Percentage of participants | 47.4 [27.4 to 68.0] | 13.3 [4.7 to 28.0] | 0.0 [0.0 to 63.2] | 13.3 [2.4 to 36.3]

ADVERSE EVENTS:
Time Frame: From start of test drug to 30 days after the last test drug intake, assessed up to 2 years after the last participant's first treatment or the last participant dies (whichever occurs first), with an average of 15 weeks for individual participant
Arm/Group | Copanlisib (Aliqopa, BAY80-6946)
All-Cause Mortality (participants affected / at risk) | 53/67
Serious Adverse Events (participants affected / at risk) | 44/67
Other Adverse Events (participants affected / at risk) | 64/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib (Aliqopa, BAY80-6946) (N=67)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Sudden death (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 9 (9)
Cystitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Splenic infection fungal (Infections and infestations) | 1 (1)
Hepatic infection fungal (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copanlisib (Aliqopa, BAY80-6946) (N=67)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Tachycardia (Cardiac disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 25 (38)
Mouth ulceration (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 20 (23)
Stomatitis (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 12 (13)
Paraesthesia oral (Gastrointestinal disorders) | 3 (5)
Asthenia (General disorders) | 3 (3)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 3 (3)
Fatigue (General disorders) | 18 (19)
Mucosal inflammation (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 7 (7)
Pyrexia (General disorders) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Lipase increased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 5 (5)
Weight decreased (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (27)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 10 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Dizziness (Nervous system disorders) | 4 (6)
Headache (Nervous system disorders) | 9 (9)
Paraesthesia (Nervous system disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 9 (10)
Haematoma (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 27 (42)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less